CLINICAL TRIAL: NCT05070910
Title: Determining the Efficacy of the Neurodevelopmental Treatment Contemporary Practice Model for the Treatment of Children With Cerebral Palsy or Other Neuromuscular Conditions to Improve Functional Outcomes.
Brief Title: NDT Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/04/10
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy; Neuromuscular Diseases; Neurodevelopment Treatment
MeSH Terms: conditions — Cerebral Palsy; Neuromuscular Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDT (Experimental): Therapy will be provided 2 days to 4 days per week for one-hour sessions
  Interventions: Behavioral: Therapy

INTERVENTIONS:
Behavioral: Therapy — The intervention performed in the practicum will not be able to be influenced by the study investigators and the intervention may be different for each child based on their needs

SUMMARY:
The purpose of this study is to determine whether there is a functional change in children with Cerebral Palsy (CP) and other neuromuscular disorders participating in Neurodevelopmental Treatment (NDT) intervention using the contemporary practice model (CPM).

ELIGIBILITY:
Inclusion Criteria:

* The children will be aged 2 to 15 years with a diagnosis of CP, hypotonia, global developmental delay and/ or neuromuscular disorders not otherwise specified.
* Children must also be willing to receive physical guidance for movement and clearly attempt to respond to simple instructions on request.
* Children and their families are available and willing to attend the practicum portion of the course for both blocks.

Exclusion Criteria:

* Parent/Guardian unable to complete the 4 required interview sessions.
* Unable to commit to attending 75% of practicum sessions.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Significant increase in functional outcomes in COPM scores | Significant change after an 8 week NDT-CPM treatment occurring from November 2, 2021 to completion on March 12, 2022
  Change functional outcomes in COPM scores after NDT-CPM treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Puyallup, Washington, United States